CLINICAL TRIAL: NCT05415709
Title: Randomized Phase I Study Assessing the Safety and Tolerability Hyperthermic Intraperitoneal Chemotherapy (HIPEC) at Completion of Interval Cytoreductive Surgery Compared to Surgery and Chemotherapy Prior to Surgery for Patients With Stage III/IV Ovarian Cancer Undergoing Neoadjuvant Chemotherapy.
Brief Title: Hyperthermic Intraperitoneal Chemotherapy With Cisplatin During Surgery or Cisplatin Before Surgery for the Treatment of Stage III or IV Ovarian, Fallopian Tube or Peritoneal Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Floor Backes, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20277; NCI-2021-06207 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-04-05; First posted 2022-06-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Serous Adenocarcinoma; Primary Peritoneal Endometrioid Adenocarcinoma; Primary Peritoneal Serous Adenocarcinoma; Stage III Fallopian Tube Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Primary Peritoneal Cancer AJCC v8; Stage IIIA Fallopian Tube Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA Primary Peritoneal Cancer AJCC v8; Stage IIIA1 Fallopian Tube Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Fallopian Tube Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Fallopian Tube Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIB Primary Peritoneal Cancer AJCC v8; Stage IIIC Fallopian Tube Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Primary Peritoneal Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8; Stage IVA Fallopian Tube Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Primary Peritoneal Cancer AJCC v8; Stage IVB Fallopian Tube Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Primary Peritoneal Cancer AJCC v8
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy; Paclitaxel; Taxes; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (carboplatin, paclitaxel, CRS, cisplatin) (Experimental): OUTLINE:
  Patients receive carboplatin IV and paclitaxel IV on day 1. Treatment repeats every 3 weeks for 3-4 cycles in the absence of disease progression or unacceptable toxicity. Within 3-4 weeks following the third or fourth neoadjuvant cycle, patients who achieve complete or partial response undergo interval cytoreductive surgery (CRS)
  Patients are randomized to 1 of 2 arms.
  ARM II: Patients receive cisplatin IV the day prior to CRS Patients undergo stool sample collection and diagnostic imaging throughout the trial.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Procedure: Cytoreductive Surgery; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Biospecimen Collection; Procedure: Diagnostic Imaging
- Arm II (carboplatin, paclitaxel, CRS, HIPEC, cisplatin) (Experimental): OUTLINE:
  Patients receive carboplatin IV and paclitaxel IV on day 1. Treatment repeats every 3 weeks for 3-4 cycles in the absence of disease progression or unacceptable toxicity. Within 3-4 weeks following the third or fourth neoadjuvant cycle, patients who achieve complete or partial response undergo interval cytoreductive surgery (CRS)
  Patients are randomized to 1 of 2 arms.
  ARM II: Patients undergo HIPEC and receive cisplatin IV over 90 minutes at the time of CRS Patients undergo stool sample collection and diagnostic imaging throughout the trial.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Procedure: Cytoreductive Surgery; Drug: Hyperthermic Intraperitoneal Chemotherapy; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Biospecimen Collection; Procedure: Diagnostic Imaging

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Cytoreductive Surgery — Undergo CRS
  Other Names: Cytoreduction
Drug: Hyperthermic Intraperitoneal Chemotherapy — Undergo HIPEC
  Other Names: HIPEC
  Arms: Arm II (carboplatin, paclitaxel, CRS, HIPEC, cisplatin)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Biospecimen Collection — Undergo stool sample collection
Procedure: Diagnostic Imaging — Undergo diagnostic imaging
  Other Names: Medical Imaging

SUMMARY:
This phase I trial studies the side effects of hyperthermic intraepithelial chemotherapy with cisplatin after surgery or cisplatin before surgery in treating patients with stage III or IV ovarian, fallopian tube or peritoneal cancer receiving chemotherapy before surgery. Hyperthermic intraepithelial chemotherapy involves the infusion of heated cytotoxic chemotherapy that circulates into the abdominal cavity at the time of surgery. Chemotherapy drugs, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving hyperthermic intraepithelial chemotherapy with cisplatin after surgery or cisplatin before surgery may kill more tumor cells compared to usual care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of intravenous (IV) cisplatin on the day prior to interval cytoreductive surgery (CRS) to administration of hyperthermic intraepithelial chemotherapy (HIPEC) with cisplatin at the completion of interval cytoreductive surgery.

SECONDARY OBJECTIVES:

I. Feasibility of each of the treatment options. II. Treatment delays. III. Perioperative outcomes. IV. Quality of life/patient reported outcomes. V. Recurrence free survival (RFS) and overall survival (OS). VI. Changes to the gut MIcrobiome

OUTLINE:

Patients receive carboplatin IV and paclitaxel IV on day 1. Treatment repeats every 3 weeks for 3-4 cycles in the absence of disease progression or unacceptable toxicity. Within 3-4 weeks following the third or fourth neoadjuvant cycle, patients who achieve complete or partial response undergo interval debulking surgery

Patients are randomized to 1 of 2 arms.

ARM I: Patients receive cisplatin IV the day prior to interval cytoreductive surgery

ARM II: Patients undergo HIPEC and receive cisplatin IV over 90 minutes at the time of interval cytoreductive surgery

All patients undergo stool sample collection and diagnostic imaging throughout the trial.

After completion of study treatment, patients are followed up for up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand (English-speaking), and willingness to sign a written, informed consent
* Age > 18 years old
* Newly diagnosed stage III or IV epithelial (serous, mucinous, or endometrioid) ovarian, fallopian tube or peritoneal cancer diagnosed by:

  * Biopsy/histology (either by interventional radiology or laparoscopy) OR
  * Cytology; If diagnosis is based on cytology the following criteria must be met:

    * Immunohistochemistry on the block from cytology to demonstrate Mullerian origin
    * Presence of pelvic mass AND CA 125 > 200kU/I AND CA125/CEA ratio > 25 at initial diagnosis
    * Omental cake or other metastases larger than 2 cm in the upper abdomen and/or regional lymph node metastasis irrespective of size (diagnosed by computed tomography [CT]/magnetic resonance imaging [MRI], ultrasound, or laparoscopy)
* Patient planned for or currently receiving neoadjuvant chemotherapy due to the fact that optimal primary CRS was determined not to be feasible by the primary surgeon
* Patient must be planned or scheduled to undergo interval cytoreductive surgery after cycle 3-4 of neoadjuvant surgery
* Completion of three cycles of neoadjuvant chemotherapy (NACT) with standard therapy (carboplatin [area under the curve (AUC) 5-6] day [D]1 + paclitaxel [175 mg/m^2] D1 every 3 weeks)

  * Following 3-4 cycles of NACT partial or complete response
  * Following 3-4 cycles of NACT at least 50% decrease in CA-125 level between pre-cycle 1 and post-cycle 3/prior to surgery
* Fit for major surgery, American Society of Anesthesiologists (ASA )1 or ASA 2
* Eastern Cooperative Oncology Group (ECOG) performance-status score of 0-2
* Serum creatinine < 1.4 mg/dL
* Creatinine clearance > 60 ml/min (Cockcroft-Gault formula)
* White blood cell count > 3.5 x 10^9 cells/L
* Absolute neutrophil count > 1.5 kg/ul
* Platelets > 100,000/ul
* Total bilirubin within 1.5 x normal institutional limits
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal
* For quality of life assessment, baseline questionnaires should be filled in before randomization

Exclusion Criteria:

* History of breast cancer or previous malignancy within 5 years prior to inclusion, with the exception of radically excised basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Low grade serious carcinoma of the ovary or borderline ovarian tumors
* History or current diagnosis of inflammatory bowel disease
* History of allergic reactions to compounds of similar chemical or biologic composition to cisplatin, carboplatin, and paclitaxel
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
* Patients in whom an optimal or complete cytoreduction cannot be performed will be excluded at the time of surgery and be replaced

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of chemotherapy-related adverse events | 30 days from perioperative treatment
  Defined by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

SECONDARY OUTCOMES:
Feasibility of chemotherapy immediately perioperatively | 1 Day prior to surgery and 1 day of surgery
  Percentage of patients able to receive planned chemotherapy the day prior to surgery or HIPEC on day of surgery
Percentage of patients in Arm C with a treatment free interval of < 8 weeks | Up to 1 year
  Percentage of patients in Arm C with a treatment free interval of < 8 weeks
Recurrence free survival | For 3-5 years after study
  time between surgery and recurrence
Tumor response | Up to 1 year
  tumor response evaluated per clinical standards
Quality of life (QOL) assessment EORTC QLQ-C30 | Baseline up to 6 months post-treatment
  Validated quality of life assessments
Changes to the gut microbiome | Within one week of re-operative appointment, cycle 1 (each cycle is 28 days) of adjuvant chemotherapy and last cycle of adjuvant chemotherapy
  metagenomic whole-genome shotgun sequencing (mWGS)

CONTACTS AND LOCATIONS:
Overall Officials: Floor Backes, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu